CLINICAL TRIAL: NCT07289711
Title: Validation and Precision Treatment of Inflammatory Subphenotypes in Acute Respiratory Distress Syndrome: A Multicenter Cohort Study
Acronym: VATIC
Status: Recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Professor, Southeast University, China
Other Study IDs: Subphenotype Of ARDS
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARDS patients with hyperinflammatory phenotype: ARDS patients with hyperinflammatory phenotype
  Interventions: Other: ARDS Inflammatory Subphenotypes

INTERVENTIONS:
Other: ARDS Inflammatory Subphenotypes — ARDS patients with idfferent Inflammatory Subphenotypes

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a common and life-threatening condition in intensive care units, characterized by substantial biological and clinical heterogeneity. Differences in patients' inflammatory responses, baseline immune function, and organ failure patterns contribute to variability in ARDS severity, treatment response, and clinical outcomes. Precision classification of ARDS based on biological and inflammatory characteristics may therefore be essential for improving patient outcomes. Previous analyses of randomized clinical trials have identified two reproducible inflammatory subphenotypes-"hyperinflammatory" and "hypoinflammatory"-which differ in organ dysfunction profiles, clinical trajectories, and responses to treatments such as fluid management strategies, corticosteroids, and ventilatory interventions. However, key uncertainties remain, including whether these inflammatory subphenotypes can be validated in Chinese ARDS populations, how various bedside prediction models perform in identifying these subphenotypes, and whether model-based subphenotype identification can guide individualized treatment decisions. This multicenter cohort study aims to: (1) validate inflammatory subphenotypes of ARDS using latent class analysis; (2) compare the predictive performance of existing bedside models for subphenotype identification; and (3) assess whether subphenotype assignment based on prediction models can guide individualized treatment strategies, including fluid management, PEEP titration, and corticosteroid use. In addition to these primary aims, the study may include other exploratory objectives, such as evaluating subphenotype stability over time, characterizing biological pathways associated with subphenotypes, and assessing additional treatment-response patterns to support future precision ARDS management strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. ARDS requiring invasive mechanical ventilation, diagnosed according to the 2023 Global definition.
3. Onset of ARDS within 72 hours.

Exclusion Criteria:

1. Refusal of informed consent by the patient's legally authorized representative.
2. Patients expected to die within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | From inclusion to 28 days
  The proportion of patients who are died within 28 days

SECONDARY OUTCOMES:
60-day mortality | From inclusion to 60 days
  The proportion of patients who are died within 60 days
Ventilator-free days at 28 days | From inclusion to 28 days
  Days alive without endotracheal intubation and invasive mechanical ventilation
Vasopressor-free days at 28 days | From inclusion to 28 days
  Days alive without use of vasopressor

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No